CLINICAL TRIAL: NCT06132789
Title: A Randomized, Single-arm, Phase Ⅰ Clinical Trial to Evaluate the Safety of Rabies Vaccine（Human Diploid Cell）for Human Use,Freeze-dried Vaccinated With Different Immunization Schedule in People Aged 10-60 Years
Brief Title: A Clinical Trial of Rabies Vaccine（Human Diploid Cell）for Human Use,Freeze-dried in a Population Aged 10-60 Years
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ab&B Bio-tech Co., Ltd.JS (Other)
Collaborators: Hubei Provincial Center for Disease Control and Prevention (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HDCV-ZHSW-03
Record Dates: First submitted 2023-11-10; First posted 2023-11-15 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Rabies
MeSH Terms: conditions — Rabies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Essen Experimental Group (18-60 years old) (Experimental): The subjects received 1 dose of 1mL Rabies Vaccine（Human Diploid Cell）for Human Use,Freeze-dried each at day 0, 3, 7, 14 and 28, with a total of 5 doses
  Interventions: Biological: Rabies Vaccine（Human Diploid Cell）for Human Use,Freeze-dried
- Essen Experimental Group (10-17 years old) (Experimental): The subjects received 1 dose of 1mL Rabies Vaccine（Human Diploid Cell）for Human Use,Freeze-dried each at day 0, 3, 7, 14 and 28, with a total of 5 doses
  Interventions: Biological: Rabies Vaccine（Human Diploid Cell）for Human Use,Freeze-dried
- Zagreb Experimental Group (18-60 years old) (Experimental): The subjects received 2 doses of 1mL Rabies Vaccine（Human Diploid Cell）for Human Use,Freeze-dried on day 0, 1 dose on day 7 and 1 dose on day 21, a total of 4 doses.
  Interventions: Biological: Rabies Vaccine（Human Diploid Cell）for Human Use,Freeze-dried
- Zagreb Experimental Group (10-17 years old) (Experimental): The subjects received 2 doses of 1mL Rabies Vaccine（Human Diploid Cell）for Human Use,Freeze-dried on day 0, 1 dose on day 7 and 1 dose on day 21, a total of 4 doses.
  Interventions: Biological: Rabies Vaccine（Human Diploid Cell）for Human Use,Freeze-dried

INTERVENTIONS:
Biological: Rabies Vaccine（Human Diploid Cell）for Human Use,Freeze-dried — This vaccine（1.0ml） is produced by Ab&b Biotechnology Co., Ltd.JS. Subjects will receive the Rabies Vaccine（Human Diploid Cell）for Human Use,Freeze-dried vaccinated by intramuscular injection.

SUMMARY:
The safety of different immunization procedures of rabies vaccine (human diploid cells) was investigated by successive design of different age groups. The two vaccination procedures were carried out successively according to the age of the subjects from the oldest to the youngest. The first 40 subjects aged 18-60 were randomly assigned to the Essen experimental group and the Zagreb experimental group in a 1:1 ratio, all of whom received the experimental vaccine. After the observation of the third dose of vaccine for at least 7 days, the preliminary safety assessment was conducted. If the incidence of grade 3 or higher adverse events associated with the experimental vaccination did not exceed 15%, and no vaccination-related death or life-threatening serious adverse events occurred, 40 subjects aged 10-17 years old were enrolled, and 40 subjects aged 10-17 years old were randomly assigned to the Essen and Zagreb trials in a 1:1 ratio. Conduct safety studies.

Safety study: All adverse events that occurred within 30 minutes, 0-7 days, and 0-30 days after each dose were collected, as well as all serious adverse events that occurred within 6 months after the first dose. Blood and urine samples were collected before the first dose and 3 days after the first dose, and blood routine, blood biochemical and urine routine tests were performed for safety assessment.

ELIGIBILITY:
Inclusion Criteria:

* Age at enrollment ranged from 10 to 60 years；
* Subjects/subjects and their guardians voluntarily agreed to participate in the study and signed an informed consent form;
* Participants and their families are permitted to participate in study follow-up visits as required by the protocol (no long-term departure or family relocation plan)；
* Female subjects were non-pregnant or lactating (negative urine pregnancy test before vaccination) and had no plans to get pregnant within 2 months after enrollment；
* The axillary temperature was < 37.3 ° C.

Exclusion Criteria:

a Exclusion criteria for the first dose:

* A history of rabies vaccine and specific passive immune preparation injection, and a history of dog or other mammal bite/scratch within the past 1 year;
* Those who are allergic to any component of the trial vaccine, or have had previous allergies to any component of the vaccine, or have had a history of severe allergies requiring medical intervention, such as anaphylactic shock, allergic laryngeal edema, Henoch-Schonlein purpura, local allergic necrosis reaction (Arthus reaction), severe urticaria, angioedema, etc;
* Fever (axillary temperature ≥37.3 ° C) within 3 days before the first dose of vaccination, acute or chronic infectious diseases (active tuberculosis, active viral hepatitis), or acute exacerbation of a chronic disease;
* Received blood/blood-related products or immune globulin within 3 months before the first dose of vaccine, or plan to use such a product after enrollment until 1 month after the last dose of vaccine;
* Vaccinate any vaccine within 14 days before the first dose of vaccine;
* Asplenia or functional asplenia due to any condition (e.g., splenectomy);
* Have been diagnosed with congenital or acquired immunodeficiency (HIV), or have been on immunosuppressive therapy within 3 months (e.g., long-term use of systemic glucocorticoids for ≥14 days at a dose of ≥2mg/kg/ day or ≥20mg/ day of prednisone or prednisone equivalent);
* Severe congenital malformations or autoimmune (hereditary) diseases, severe chronic diseases (including but not limited to thalassemia, heart disease, kidney disease, diabetes mellitus, hereditary allergies, Guillain-Barre syndrome, etc.);
* People with a medical or family history of seizures, epilepsy, encephalopathy and psychosis;
* Contraindications to intramuscular injection (e.g. having been diagnosed with thrombocytopenia, any coagulopathy, or receiving anticoagulant therapy);
* Drug-uncontrolled hypertension, defined as pre-enrollment systolic blood pressure ≥160mmHg and/or diastolic blood pressure ≥100mmHg (for adults aged 18 years and over);
* Are participating in other investigational or unregistered clinical studies of products (drugs or vaccines), or plan to participate in other clinical studies before the end of this clinical study;
* Patients with clinically significant abnormalities in laboratory tests such as blood routine, blood biochemistry, and urine routine could not be enrolled according to the comprehensive judgment of the investigators;
* The investigator considered the subject to have any condition that might interfere with the assessment of the purpose of the study.

b Exclusion criteria for subsequent doses:

* Positive urine pregnancy test；
* Severe anaphylaxis after the previous dose;
* Grade 4 adverse events associated with trial vaccination after the previous dose;
* Exposure during the course (bite or scratch from dogs, cats or other mammals);
* Subject has any other conditions that warrant discontinuation of vaccination as determined by the investigator.

Ages: 10 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 80 (Actual)
Dates: Start 2023-11-27 (Actual); Primary Completion 2024-08-16 (Actual); Study Completion 2024-08-16 (Actual)

PRIMARY OUTCOMES:
The occurrence of adverse events/reactions within 1 month from the first dose to full immunization; | Within 1 month from the first dose to full immunization
  The occurrence of adverse events/reactions within 1 month from the first dose to full immunization;
The occurrence of serious adverse events/reactions within 6 month from the first dose to full immunization; | Within 6 month from the first dose to full immunization
  The occurrence of serious adverse events/reactions within 6 month from the first dose to full immunization;
The abnormal occurrence of laboratory indicators (blood biochemistry, blood routine and urine routine) 3 days after the first dose of vaccination | 3 days after the first dose
  The abnormal occurrence of laboratory indicators (blood biochemistry, blood routine and urine routine) 3 days after the first dose of vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Xianfeng Zhang, Master, Principal Investigator — Hubei Provincial Center for Disease Control and Prevention
Locations (1):
- Gucheng Center for Disease Control and Prevention, Xiangyang, Hubei, China

IPD SHARING:
Plan to Share IPD: No